CLINICAL TRIAL: NCT06178952
Title: Transcranial Pulse Stimulation (TPS) in Post-COVID-19
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Roland Beisteiner, Professor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 102307161; 102307161 (Other: BASG (Austrian Agency for Health and Food Safety))
Record Dates: First submitted 2023-12-20; First posted 2023-12-21 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Post-COVID-19 Syndrome; Fatigue
Keywords: Transcranial Pulse Stimulation; Post-COVID-19; Fatigue; Non-invasive brain stimulation
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue

STUDY DESIGN:
Intervention Model Description: Prospective, double-blind, randomized, parallel group, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants as well as the principal investigator, evaluating investigators, and the teams responsible for conducting stimulations, neuropsychological testing, and MR testing will be blinded. Specific individuals responsible for the organization of the study, who are neither involved in stimulation nor data collection, will not be blinded and will apply the verum or sham standoff device to the NEUROLITH system for a specific patient. As the stimulation team members won't have knowledge of the standoff device in use, they will remain completely blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Verum TPS (Experimental): Participants will receive 5 Verum TPS sessions over a period of 10 days, with a singular daily session, each lasting approximately 30 minutes
  Interventions: Device: Transcranial pulse stimulation Verum
- Sham TPS (Sham Comparator): Participants will receive 5 Sham TPS sessions over a period of 10 days, with a singular daily session, each lasting approximately 30 minutes
  Interventions: Device: Transcranial pulse stimulation Sham

INTERVENTIONS:
Device: Transcranial pulse stimulation Verum — Participants are slated to undergo a total of five TPS sessions over a 10-day interval. Each stimulation session will endure approximately 30 minutes and will be administered once daily.
  Arms: Verum TPS
Device: Transcranial pulse stimulation Sham — Placebo treatment will be performed using the same medical device, handpiece and treatment paradigm as in the verum treatment with one difference: the standoff device at the end of the handpiece. This device is designed to replicate the appearance, feel, and sound of the verum system, while omitting the transmission of any pulses.
  Arms: Sham TPS

SUMMARY:
The objective of the present study is to demonstrate treatment efficacy of transcranial pulse stimulation for patients with Post-COVID-19 related neurological symptoms (fatigue, cognitive deficits, mood deterioration). Fatigue, as measured by the Fatigue Impact Scale (FIS), will represent the primary outcome variable. The verum treatment will be compared to a sham (placebo) condition.

DETAILED DESCRIPTION:
This clinical trial aims to investigate the treatment efficacy of transcranial pulse stimulation (TPS) using the NEUROLITH device (Storz Medical AG, Tägerwilen, Switzerland) in individuals with neurological post-COVID-19-symptoms. TPS is a novel brain stimulation therapy based on non-invasive ultrasound pulses and first published in 2019 by the Medical University of Vienna, Austria (Beisteiner et al. Advanced Science, 2019). The study employs a double-blind, randomized, placebo-controlled design with parallel groups (verum vs. sham). The anticipated timeframe for the entire study is 2 years, during which each participant is expected to be actively engaged for a period of 3-4 months. The aim is to include 102 patients. The randomization ratio is 1:1, ensuring an even distribution between the verum (active treatment) and sham (placebo) groups. Three assessment points are scheduled (Baseline, PostStim, 1monthPostStim). Furthermore, to determine potential effects over time, limited data collection (involving only FIS, BDI-II, SF-36 and BI-PEM) is planned at later time points, specifically at 3 months post-stimulation, 6 months post-stimulation, 12 months post-stimulation, and 24 months post-stimulation.

Hypotheses

* H0: There is no significant difference in the effectiveness of transcranial pulse stimulation (TPS) and placebo treatment in improving primary and secondary endpoints.
* H1: There is a significant difference in the effectiveness of transcranial pulse stimulation (TPS) and placebo treatment in improving primary and secondary endpoints.

Timeline

Each study participant will undergo the following sequence:

1. Initial information session and clarification of relevant medical findings regarding inclusion and exclusion criteria
2. Baseline screening:

   * 3-4 assessment sessions per patient within 14 days, including informed consent
   * Patients who do not meet the predefined cut-off values for BDI, FIS, and MoCA will be excluded from subsequent study phases
3. Transcranial pulse stimulation

   * 5 stimulations per patient within 10 days
   * One stimulation per day lasting approximately 30 minutes.
4. Post-stimulation assessment (PostStim)

   * Conducted during the week following brain stimulation
   * 2-3 assessment sessions per patient within 7 days
5. One-month post-stimulation assessment (1monthPostStim)

   * Conducted one month after brain stimulation
   * 2-3 assessment sessions per patient within 7 days

Deviations of + 5 days from the intended timeline are considered tolerable.

Sample Size Calculation

The sample size calculation conducted with G*Power incorporated a small effect size (f = .10), α error probability of .05, and a power of 0.8, resulting in an estimate of 102 patients.

Important note: Originally, the study was designed as a multicenter study with the still-existing Austrian center (N=90) and an Italian center (N=30). Since study realization at the Italian center was ultimately not possible, the trial was streamlined to a single-center design. Consequently, enrollment at the Austrian center was refined so that at least 102 participants would reach the primary endpoint, thus meeting the original sample-size requirement. This administrative change was made prior to any analyses and does not affect the prespecified endpoints or procedures.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* PCR-confirmed SARS-CoV-2 infection, laboratory confirmed antibody detection for SARS-CoV-2, or physician-verified COVID-19 infection
* At least 12 months after initial SARS-CoV-2 infection that led to Post-COVID (subsequent SARS-CoV-2 infections are not a reason for exclusion)
* Diagnosis of Post-COVID Syndrome or independent suspected diagnosis of Post-COVID Syndrome (Considering that physicians generally hesitate to provide clear-cut Post-COVID diagnoses, a tentative diagnosis by an independent general practitioner or a specialist in a field associated with Post-COVID will suffice for entering this study)
* Age: 20-80
* Evidence of a negative pregnancy test if medically adequate

Exclusion Criteria:

* Clinically relevant realization of pre-COVID diseases with similar symptoms as Post-COVID
* MoCA score <17 (cut-off for dementia)
* BDI-II score ≥29 (cut-off for severe depression)
* FIS <10 (cut-off for no fatigue)
* Brain implants
* Non-MR-compatible metal parts in the body
* Metal parts in the head
* Use of anticoagulants
* Non-MR-compatible claustrophobia
* Non-MR-compatible pacemaker
* Pregnant and breastfeeding women
* Clinically relevant history of surgery on the head, heart, or vessels
* Relevant corticosteroid treatments administered within 6 weeks prior to the first application
* Tumor of the head if relevant for treatment
* Blood clotting disorders
* Participation in other studies

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue Impact Scale (FIS) | Baseline - 1 week after stimulation - 1 month after stimulation
  The Fatigue Impact Scale (Fisk et al., 1994) is an instrument to measure the impact of fatigue symptoms. This self-report measure consists of 40 items divided into three subscales: cognitive functioning (10 items), physical functioning (10 items) and psychosocial functioning (20 items). In the validated German version, the statements are scored from 0-4 (0=never, 4=very often) leading to a total score of 0-160.

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI-II) | Baseline - 1 week after stimulation - 1 month after stimulation
  The Beck Depression Inventory (BDI-II) is one of the most widely used instruments for measuring the severity of depression. It is a 21-item questionnaire for self-evaluation with 0-3 scores per item, ranging from 0 (normal state) to 63 (severe depression).
Montreal Cognitive Assessment (MOCA) | Baseline - 1 week after stimulation - 1 month after stimulation
  Montreal Cognitive Assessment (Nasreddine et al., 2005) is a clinical standard test for evaluating the following cognitive functions: visuospatial/executive, naming, memory, attention, language, abstraction, recall and orientation. The maximum score is 30 points.
36-Item Short Form Health Survey (SF-36) | Baseline - 1 week after stimulation - 1 month after stimulation
  The 36-item short-form health survey (Ware et al., 1992) is a widely used instrument to measure quality of life. The 36-item patient-reported survey covers eight health concepts including physical functioning (10 items), role limitations due to physical health (4 items), role limitations due to emotional problems (3 items), energy/fatigue (4 items), emotional well-being (5 items), social functioning (2 items), pain (2 items), and general health (5 items). All questions are scored on a scale from 0 (worst health) to 100 (best health).
Trail Making Test A and B (TMT-A and TMT-B) | Baseline - 1 week after stimulation - 1 month after stimulation
  The Trail Making Test (Reitan et al., 1958) consist of two parts A and B. For each part, patients need to fulfill a task by connecting letters and/or numbers in the right way. The scoring of both parts is done by taking the time required to complete them.
Positive and Negative Affect Schedule (PANAS) | Baseline - 1 week after stimulation - 1 month after stimulation
  The Positive and Negative Affect Schedule (Watson et al., 1988) is an instrument to assess mood, specifically distinguishing between positive and negative affect. It has two subscales (positive and negative) and consists out of 20 items which are scored using a 5-point scale (1= not at all - 5 = extremely).
Beck Anxiety Inventory (BAI) | Baseline - 1 week after stimulation - 1 month after stimulation
  The Beck Anxiety Inventory (Beck et al., 1988) is a self-reported scale to measure anxiety. It consists of 21 items, which are scored from 0-3. The BAI has a total range from 0 to 63.
Six Minute Walking Test (6MWT) | Baseline - 1 week after stimulation - 1 month after stimulation
  The six-minute walking test, developed by the American Thoracic Society 2002, is an exercise test to assess aerobic capacity and endurance. The patients are asked to walk as far as they can within 6 minutes. Subjective tests (Borg-Scale, 0-10) will be administers before and after walking.
Test of Attentional Performance (TAP) | Baseline - 1 week after stimulation - 1 month after stimulation
  The Test of Attentional Performance (Zimmermann et al., 2002) is an instrument to measure attentional function. There are 14 subscales, including Sustained Attention, Vigilance, and Divided Attention. It will be carried out digitally using the TAP software package.
Verbal Learning and Memory Test (VLMT) | Baseline - 1 week after stimulation - 1 month after stimulation
  The German version of the Verbal Learning Memory Test by Helmstaedter and colleagues (2001) is an instrument to measure different parameters of declarative verbal memory such as learning or recognition performance. It consists of a learning phase, in which patients need to learn two lists of 15 words each, a delayed recall and a recognition test.
Stroop color word test (STROOP) | Baseline - 1 week after stimulation - 1 month after stimulation
  The Stroop Color-Word Test (Stroop, 1935) is a useful and reliable psychological assessment tool (Lezak, Howieson, & Loring, 2004) that measures a person's ability to inhibit an automatic response in favor of an atypical one. Specifically, it involves identifying the ink color of incongruously labeled color words (van Boxtel et al., 2001). The test can measure cognitive performance functions such as naming speed, selectivity, and alertness (Bäumler & Stroop, 1985).
Satisfaction With Life Scale (SWLS) | Baseline - 1 week after stimulation - 1 month after stimulation
  The SWLS (Satisfaction with Life Scale), developed by Diener and colleagues (1985), is a widely used self-report questionnaire designed to measure individuals' subjective satisfaction with their own lives. It consists of five items that capture different aspects of life satisfaction.
Somatization subscale of the Symptom Check List-90-R (SCL-90-R SOM) | Baseline - 1 week after stimulation - 1 month after stimulation
  The SCL-90-R (Schmitz et al., 2000) is a 90-item self-report symptom inventory used in clinical and research settings to evaluate psychological symptoms and distress. Only the SOM (Somatization) subscale within the SCL-90-R will be used for the present study. It consists of 12 items on a 5-point Likert scale that assess physical symptoms. The maximum score for the subscale is 48 points.
Post-Exertional Malaise (BI-PEM) | Baseline - 1 week after stimulation - 1 month after stimulation
  The German version of the DSQ PEM questionnaire (Cotler et al., 2018; Jason & Sunnquist, 2018) comprises three subscales and a total of 11 items, focusing on post-exertional malaise. The subscales include questions concerning frequency, severity and duration of the symptoms after engaging in activities over the past 6 months.
Neuroimaging | Baseline - 1 week after stimulation - 1 month after stimulation
  Magnetic resonance imaging (MRI) will be recorded the week before, the week after and 1 month after TPS stimulations by center 1 (Vienna) for the Austrian study population. MR measurements will be performed using a 3 T SIEMENS PRISMA MR with a 64-channel head coil. MRI images will be obtained to assess changes in structural and functional brain connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Beisteiner, Prof., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the medical information used in the study, access to individual data will not be provided to other researchers.

REFERENCES:
- [Background] Beisteiner R, Matt E, Fan C, Baldysiak H, Schonfeld M, Philippi Novak T, Amini A, Aslan T, Reinecke R, Lehrner J, Weber A, Reime U, Goldenstedt C, Marlinghaus E, Hallett M, Lohse-Busch H. Transcranial Pulse Stimulation with Ultrasound in Alzheimer's Disease-A New Navigated Focal Brain Therapy. Adv Sci (Weinh). 2019 Dec 23;7(3):1902583. doi: 10.1002/advs.201902583. eCollection 2020 Feb. PMID 32042569
- [Background] Beisteiner R, Hallett M, Lozano AM. Ultrasound Neuromodulation as a New Brain Therapy. Adv Sci (Weinh). 2023 May;10(14):e2205634. doi: 10.1002/advs.202205634. Epub 2023 Mar 24. PMID 36961104
- [Background] Cont C, Stute N, Galli A, Schulte C, Logmin K, Trenado C, Wojtecki L. Retrospective real-world pilot data on transcranial pulse stimulation in mild to severe Alzheimer's patients. Front Neurol. 2022 Sep 14;13:948204. doi: 10.3389/fneur.2022.948204. eCollection 2022. PMID 36188380
- [Background] Douaud G, Lee S, Alfaro-Almagro F, Arthofer C, Wang C, McCarthy P, Lange F, Andersson JLR, Griffanti L, Duff E, Jbabdi S, Taschler B, Keating P, Winkler AM, Collins R, Matthews PM, Allen N, Miller KL, Nichols TE, Smith SM. SARS-CoV-2 is associated with changes in brain structure in UK Biobank. Nature. 2022 Apr;604(7907):697-707. doi: 10.1038/s41586-022-04569-5. Epub 2022 Mar 7. PMID 35255491
- [Background] Ashraf N, Abou Shaar B, Taha RM, Arabi TZ, Sabbah BN, Alkodaymi MS, Omrani OA, Makhzoum T, Almahfoudh NE, Al-Hammad QA, Hejazi W, Obeidat Y, Osman N, Al-Kattan KM, Berbari EF, Tleyjeh IM. A systematic review of trials currently investigating therapeutic modalities for post-acute COVID-19 syndrome and registered on WHO International Clinical Trials Platform. Clin Microbiol Infect. 2023 May;29(5):570-577. doi: 10.1016/j.cmi.2023.01.007. Epub 2023 Jan 13. PMID 36642173
- [Background] Han Q, Zheng B, Daines L, Sheikh A. Long-Term Sequelae of COVID-19: A Systematic Review and Meta-Analysis of One-Year Follow-Up Studies on Post-COVID Symptoms. Pathogens. 2022 Feb 19;11(2):269. doi: 10.3390/pathogens11020269. PMID 35215212
- [Background] Kubota T, Kuroda N, Sone D. Neuropsychiatric aspects of long COVID: A comprehensive review. Psychiatry Clin Neurosci. 2023 Feb;77(2):84-93. doi: 10.1111/pcn.13508. Epub 2022 Dec 12. PMID 36385449
- [Background] Linnhoff S, Koehler L, Haghikia A, Zaehle T. The therapeutic potential of non-invasive brain stimulation for the treatment of Long-COVID-related cognitive fatigue. Front Immunol. 2023 Jan 9;13:935614. doi: 10.3389/fimmu.2022.935614. eCollection 2022. PMID 36700201
- [Background] Matt E, Kaindl L, Tenk S, Egger A, Kolarova T, Karahasanovic N, Amini A, Arslan A, Saricicek K, Weber A, Beisteiner R. First evidence of long-term effects of transcranial pulse stimulation (TPS) on the human brain. J Transl Med. 2022 Jan 15;20(1):26. doi: 10.1186/s12967-021-03222-5. PMID 35033118
- [Background] Matt E, Dorl G, Beisteiner R. Transcranial pulse stimulation (TPS) improves depression in AD patients on state-of-the-art treatment. Alzheimers Dement (N Y). 2022 Feb 10;8(1):e12245. doi: 10.1002/trc2.12245. eCollection 2022. PMID 35169611
- [Background] O'Sullivan O. Long-term sequelae following previous coronavirus epidemics. Clin Med (Lond). 2021 Jan;21(1):e68-e70. doi: 10.7861/clinmed.2020-0204. Epub 2020 Nov 3. PMID 33144403
- [Background] Pinzon RT, Wijaya VO, Jody AA, Nunsio PN, Buana RB. Persistent neurological manifestations in long COVID-19 syndrome: A systematic review and meta-analysis. J Infect Public Health. 2022 Aug;15(8):856-869. doi: 10.1016/j.jiph.2022.06.013. Epub 2022 Jun 23. PMID 35785594
- [Background] Popescu T, Pernet C, Beisteiner R. Transcranial ultrasound pulse stimulation reduces cortical atrophy in Alzheimer's patients: A follow-up study. Alzheimers Dement (N Y). 2021 Feb 25;7(1):e12121. doi: 10.1002/trc2.12121. eCollection 2021. PMID 33681449
- [Background] Radjenovic S, Dorl G, Gaal M, Beisteiner R. Safety of Clinical Ultrasound Neuromodulation. Brain Sci. 2022 Sep 22;12(10):1277. doi: 10.3390/brainsci12101277. PMID 36291211
- [Background] Santana K, Franca E, Sato J, Silva A, Queiroz M, de Farias J, Rodrigues D, Souza I, Ribeiro V, Caparelli-Daquer E, Teixeira AL, Charvet L, Datta A, Bikson M, Andrade S. Non-invasive brain stimulation for fatigue in post-acute sequelae of SARS-CoV-2 (PASC). Brain Stimul. 2023 Jan-Feb;16(1):100-107. doi: 10.1016/j.brs.2023.01.1672. Epub 2023 Jan 21. PMID 36693536
- [Background] Soriano JB, Murthy S, Marshall JC, Relan P, Diaz JV; WHO Clinical Case Definition Working Group on Post-COVID-19 Condition. A clinical case definition of post-COVID-19 condition by a Delphi consensus. Lancet Infect Dis. 2022 Apr;22(4):e102-e107. doi: 10.1016/S1473-3099(21)00703-9. Epub 2021 Dec 21. PMID 34951953
- [Background] Tran VT, Porcher R, Pane I, Ravaud P. Course of post COVID-19 disease symptoms over time in the ComPaRe long COVID prospective e-cohort. Nat Commun. 2022 Apr 5;13(1):1812. doi: 10.1038/s41467-022-29513-z. PMID 35383197
- [Background] Weinreb E, Moses E. Mechanistic insights into ultrasonic neurostimulation of disconnected neurons using single short pulses. Brain Stimul. 2022 May-Jun;15(3):769-779. doi: 10.1016/j.brs.2022.05.004. Epub 2022 May 11. PMID 35561960
- [Background] Zeng N, Zhao YM, Yan W, Li C, Lu QD, Liu L, Ni SY, Mei H, Yuan K, Shi L, Li P, Fan TT, Yuan JL, Vitiello MV, Kosten T, Kondratiuk AL, Sun HQ, Tang XD, Liu MY, Lalvani A, Shi J, Bao YP, Lu L. A systematic review and meta-analysis of long term physical and mental sequelae of COVID-19 pandemic: call for research priority and action. Mol Psychiatry. 2023 Jan;28(1):423-433. doi: 10.1038/s41380-022-01614-7. Epub 2022 Jun 6. PMID 35668159